CLINICAL TRIAL: NCT03814616
Title: A Randomized, Open-Label Exploratory Study To Determine The Efficacy Of Different Treatment Regimens Of Pyramax® (Pyronaridine-Artesunate) In Asymptomatic Carriers Of Plasmodium Falciparum Monoinfections
Brief Title: Pyramax in Asymptomatic Carriers of P. Falciparum Monoinfections
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP-C-026-18
Record Dates: First submitted 2018-09-13; First posted 2019-01-24 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Malaria,Falciparum
Keywords: Asymptomatic malaria
MeSH Terms: conditions — Malaria, Falciparum | interventions — pyronaridine; Artesunate; pyronaridine tetraphosphate, artesunate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm Pyramax 3 days (Experimental): Pyramax (pyronaridine tetraphosphate 180mg:artesunate 60mg) will be administered, once per day according to body weight for three days (Arm A)
  Interventions: Drug: Pyronaridine tetraphosphate 180mg:artesunate 60mg
- Arm Pyramax 2 days (Experimental): Pyramax (pyronaridine tetraphosphate 180mg:artesunate 60mg) will be administered, once per day according to body weight for two days (Arm B)
  Interventions: Drug: Pyronaridine tetraphosphate 180mg:artesunate 60mg
- Arm Pyramax 1 day (Experimental): Pyramax (pyronaridine tetraphosphate 180mg:artesunate 60mg) will be administered, once per day according to body weight for one day (Arm C)
  Interventions: Drug: Pyronaridine tetraphosphate 180mg:artesunate 60mg

INTERVENTIONS:
Drug: Pyronaridine tetraphosphate 180mg:artesunate 60mg — ACT
  Other Names: Pyramax

SUMMARY:
This study will assess the efficacy of Pyramax administered for three-day, two-day or one day, in clearing a P. falciparum infection in asymptomatic carriers.

.

DETAILED DESCRIPTION:
This is a randomized, open-label, three-arm, out-patient study in asymptomatic individuals with P. falciparum monoinfection confirmed at baseline, who are >5 years of age and >20kg body weight. A total of 300 participants will be randomised into the study; 100 participants in each of three treatment arms.

Patients who fulfil the entry criteria (all inclusion and none of the exclusion criteria) will be recruited and randomized to receive Pyramax orally for three days, two days or one day in a randomization ratio of 1:1:1.

All participants will be followed until Day 63 (counted from day 0) and blood samples will be taken on Days 0, 1, 2, 3, 7, 14, 21, 28, 35, 42 and 63 for malaria diagnostics, parasite density and qPCR. In addition, blood samples reverse-transcriptase (RT)-PCR will be taken on Days 0, 1, 2, 3, 7 and 14.

Participants will be administered local SOC treatment if they meet any of the protocol-specific criteria of treatment failure: Early treatment failure, Late clinical failure, or Late parasitological failure up to and including Day 63, or if the participant withdraws at any time before Day 63, and is parasite positive.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of asymptomatic infection with Plasmodium falciparum monoinfection on thin and thick blood smears with parasite density between 20/µL and 50,000/µL
2. Absence of any clinical symptoms of malaria at the time of enrolment and within 72 hours before enrolment
3. Age >5 years old and >20 kg body weight
4. Ability to swallow oral medication
5. Evidence of a personally signed and dated Informed Consent document indicating that the participant (or a legally acceptable representative if a participant is <18 years of age) has been informed of all pertinent aspects of the study and that all questions by the participant have been sufficiently answered. Assent will be obtained from participants <18 years of age as required by national regulations.
6. Participants who are willing to and are able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Haemoglobin <7 g/dL (measured at screening)
2. History of having received any antimalarial treatment (alone or in combination) during the following periods before screening:

   1. Piperaquine, mefloquine, naphthoquine or sulfadoxine-pyrimethamine within 6 weeks prior to screening
   2. Amodiaquine, chloroquine within 4 weeks prior to screening
   3. Any artemisinin derivative (artesunate, artemether or dihydroartemisinin), quinine, lumefantrine or any other anti-malarial treatment or antibiotic with antimalarial activity (including cotrimoxazole, tetracyclines, quinolones and fluoroquinolones and azithromycin) within 14 days prior to screening
3. Any herbal products or traditional medicines during the 7 days prior to screening (if spontaneously reported by the patient)
4. Known allergy to the study drugs (pyronaridine and/or any artemisinin derivatives)
5. Positive urinary pregnancy test for women of reproductive age
6. Lactating women
7. Evidence of severe malnutrition
8. Participation in other studies within 30 days before the current study begins and/or during study participation
9. Inability to comprehend and/or unwillingness to follow the study protocol
10. Previously randomized in this study
11. Severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study. Examples would include but not limited to:

    1. Immunological disorders (including known seropositive HIV antibody),
    2. Severe psychiatric disorders (active depression, recent history of depression, generalised anxiety, psychosis, schizophrenia or other major psychiatric disorders) and major medical disorders related to cardiovascular, respiratory (including active tuberculosis), renal, gastrointestinal, endocrine, infectious, malignancy, neurological (including auditory) and history of convulsions or other abnormality (including recent head trauma),
    3. Clinical signs or symptoms of hepatic injury (such as nausea, abdominal pain associated with jaundice) or known severe liver disease (i.e. decompensated cirrhosis, Child-Pugh stage 3 or 4)
12. Participant the Investigator considers at particular risk of receiving an anti-malarial or of participating in the study

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
PCR-adjusted APR at Day 28 (based on slide assessment by microscopy) | Day 28
  To assess the efficacy of each dosing regimen PCR-adjusted Adequate parasitological response (APR) at Day 28

SECONDARY OUTCOMES:
PCR-adjusted APR | 63 days
  To assess the efficacy of each dosing regimen PCR-adjusted APR at Day 63
PCR-unadjusted APR | 63 days
  To assess the efficacy of each dosing regimen PCR-unadjusted APR at Day 63
Rate of recurrent infections, recrudescence and new infections | 63 days
  To assess the efficacy of each dosing regimen on rate of recurrent infections, recrudescence and new infections
Proportion of parasite free participants | 4 days
  Proportion of participants who are parasite free by 4-8 hours, Day 1, Day 2 and Day 3 post first dosing
Gametocyte incidence | 14 days
  The area under the curve (AUC) up to Day 14 (post first dose) of gametocytes in participants with gametocytes at baseline, and separately in participants without gametocytes at baseline
Adverse Events | 63 days
  * Number (%) of patients and number of events with:
    * TEAEs,
    * serious TEAEs,
    * study drug related TEAEs,
    * study drug related serious TEAEs,
    * malaria-related TEAEs,
    * malaria-related serious TEAEs
  * Number (%) of patients with TEAEs and drug-related TEAEs by maximum severity, based on Grade 1 to Grade 5 (CTCAE V4.03) severity grading Adverse events will be coded by MedDRA primary system organ class and preferred term.
  * Hepatotoxicity related TEAEs o The number and percentage of patients with hepatotoxicity related TEAEs, based on the Standard MedDRA Query (SMQ) narrow search "Drug-related hepatic disorders" will be summarised and clinical biochemistry parameters
Clinical laboratory data - Haematology | 63 days
  Haemoglobin, haematocrit, erythrocytes, platelets, white blood cells, neutrophils, lymphocytes, monocytes, eosinophils, basophils will be summarised over time, as absolute values and changes from baseline with the number of observations, mean, standard deviation, median, quartiles, minimum and maximum. SI units will be used to summarise the data.
Clinical laboratory data - Biochemistry | 63 days
  Total and conjugated bilirubin will be summarised over time, as absolute values and changes from baseline with the number of observations, mean, standard deviation, median, quartiles, minimum and maximum. SI units will be used to summarise the data.
Clinical laboratory data - Liver Enzymes | 63 days
  Alanine aminotransaminase (ALT), Aspartate aminotransaminase (AST), Alkaline Phosphatase will be summarised over time, as absolute values and changes from baseline with the number of observations, mean, standard deviation, median, quartiles, minimum and maximum. IU/L units will be used to summarise the data
Clinical laboratory data - Liver Enzyme Elevations | 63 days
  The number (%) of participants with liver enzyme elevations after first drug administration as defined below will be summarised.
  * ALT or AST > 3 x Upper Limit of Normal (ULN)
  * ALT or AST > 5 x ULN
  * ALT or AST > 8 x ULN
  * ALT or AST > 3 x ULN and bilirubin > 2 x ULN at the same time point (when conjugated bilirubin fraction is missing)
  * ALT or AST > 3 x ULN and bilirubin > 2 x ULN, together with a conjugated bilirubin fraction >35% (Potential Hy's law cases), at the same time point
Vital signs - Blood pressure | 63 days
  Supine systolic and diastolic blood pressure (mm Hg) absolute values and changes from baseline will be summarised by time point with the number of observations, mean, standard deviation, median, minimum and maximum, and quartiles
Vital signs - Pulse rate | 63 days
  Pulse rate (bpm) absolute values and changes from baseline will be summarised by time point with the number of observations, mean, standard deviation, median, minimum and maximum, and quartiles
Vital signs - Temperature | 63 days
  Temperature (degrees Celsius) absolute values and changes from baseline will be summarised by time point with the number of observations, mean, standard deviation, median, minimum and maximum, and quartiles

OTHER OUTCOMES:
Parasite free by qPCR quantification | 63 days
  To estimate the proportion of participants who are parasite free by qPCR quantification.
PCR-adjusted APR by qPCR | 63 days
  To estimate PCR-adjusted APR by qPCR.To estimate PCR-unadjusted APR by qPCR. To estimate the rate of recurrent infections, recrudescences and new infections by qPCR until Day 63 (post first dose) by KM analysis.
Percentage change in gametocytaemia. | 63 days
  In participants with positive detection of gametocytes by reverse transcriptase (RT)-PCR at baseline, to evaluate percentage reduction in gametocytaemia.
AUC of gametocytaemia by RT-PCR | 14 days
  To estimate area under the curve (AUC) up to Day 14 of gametocytaemia by RT-PCR, in participants with positive RT-PCR at baseline and separately in participants with negative RT-PCR at baseline
Relationship between artesunate and pyronaridine concentration and efficacy | 28 days
  To explore the relationship between artesunate and pyronaridine concentration and efficacy (PCR-adjusted APR at Day 28, based on slide assessment by microscopy)

CONTACTS AND LOCATIONS:
Overall Officials: Jang Sik Shin, Study Director — Shin Poong
Locations (2):
- MRC Unit The Gambia at the London School of Hygiene and Tropical Medicine,, Fajara, City of Banjul, The Gambia
- Tropical Diseases Research Centre, Ndola, Zambia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dabira ED, Hachizovu S, Conteh B, Mendy A, Nyang H, Lawal B, Ndiath MO, Mulenga JM, Mwanza S, Borghini-Fuhrer I, Arbe-Barnes S, Miller R, Shin J, Duparc S, D'Alessandro U, Manyando C, Achan J. Efficacy, Safety and Tolerability of Pyronaridine-artesunate in Asymptomatic Malaria-infected Individuals: a Randomized Controlled Trial. Clin Infect Dis. 2022 Jan 29;74(2):180-188. doi: 10.1093/cid/ciab425. PMID 33983371